CLINICAL TRIAL: NCT04848740
Title: Human Fresh Corneal Lenticule Implantation Criteria in Progressive Corneal Disease Using Relex-Smile
Acronym: Relex-Smile
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeHPristina1
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Progressive Disease of Corneae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FRESH CORNEAL LENTICULE IMPLANTATION (Other): The aim in our study is to describe the importance of stroma as criteria of corneal thickness at implanting human fresh corneal lenticule in progressive corneal disease.
  We have conclude that every biomechanical instability of corneal stroma function(abnormal increase collagen activity,decrease proteinase inhibitors,excessive premature keratocyte apoptosis) describe the role of stroma in corneal thickness.
  Interventions: Device: ReLex-smile

INTERVENTIONS:
Device: ReLex-smile — Using VisuMax femtosecond laser we created the stromal pocket with diameter of 7.6 to 8.0 mm (1 mm larger than the optical zone of the donor lenticule) and cap thickness set to 130 μm from corneal surface and 4 mm superior incision. Hinge position flap was set at 90° angle 50° and width 4 mm, side cut angle 90°. The pocket was dissected using a blunt spatula washed with normal saline. The lenticule was held with lenticule forceps and gently inserted into the pocket through the 4 mm superior incision. Incision position changed according to the position of the highest K values We noticed during intervention that implantation of fresh lenticule depends from corneal thickness, for example if c.th.is 300-400 μm we implanted 1/2 stroma, if c.th.is 400 μm or more we implanted 1/3 stroma Example: if corneal thickness is 300 μm we implanted 150 μm (becoming 450 μm) we added more stroma due to more live keratocytes and stromal steam cells, aiming to overcome dead and non-functional keratocytes

SUMMARY:
Stroma is a fibrous, tough, transparent and the thickest layer of the corneae. The stroma is composed of organised collagen, which maintains transparency. Keratocytes are located between the lamella collagen fibers and secrete an extracellular matrix, which includes collagen, proteoglycan, crystalline proteins to maintain corneal transparency.

DETAILED DESCRIPTION:
Knowing the importance of stroma(90%) in function and anatomy of corneae (transparence, curvature, strength, protection) the inner eye structures from external environment, we have examined the role and function of stroma as a main factor of corneal thickness in implanting fresh corneal lenticule in progressive corneal disease.

We have studied that in many clinical cases where the corneal epithelium and endothelium are healthy and functioning, the cornea can still lose it's transparency by different corneal stromal pathologies (infection ,keratoconus, inflammation ,neurodegeneration and corneal dystrophies).

ELIGIBILITY:
Inclusion Criteria:

* progressive corneal disease with thin corneal thickness
* corneal low transparenc
* low visual acuity

Exclusion Criteria:

* active anterior segment pathology
* previous corneal or anterior segment surgery
* other infection etc.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Increase of corneal thickness | 24 months
  Increase of corneal central thickness using human fresh corneal lenticule with stromal stem cells and live keratocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided